CLINICAL TRIAL: NCT02984358
Title: Effect of Chronic Mycoprotein Consumption, and of Its Nucleotide Content, in Uric Acid Concentrations and Other Markers of Metabolic Health in Adults
Brief Title: Chronic Mycoprotein Consumption and Nucleotide Content in Metabolic Health
Acronym: MYTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 660065613
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Animal protein based diet (Placebo Comparator): Seven day fully controlled normocaloric diet (1.2 g/ kg body weight of protein per day), with the main protein source at the two main meals (lunch and dinner) being provided by animal products (meat and fish).
  Interventions: Other: Animal protein based diet
- Low-nucleotide mycoprotein based diet (Active Comparator): Seven day fully controlled normocaloric diet (1.2 g/ kg body weight of protein per day), with the main protein source at the two main meals (lunch and dinner) being provided by nucleotide-depleted mycoprotein products (commercial Quorn products).
  Interventions: Other: Low-nucleotide mycoprotein based diet
- High-nucleotide mycoprotein based diet (Active Comparator): Seven day fully controlled normocaloric diet (1.2 g/ kg body weight of protein per day), with the main protein source at the two main meals (lunch and dinner) being provided by nucleotide-rich mycoprotein products.
  Interventions: Other: High-nucleotide mycoprotein based diet

INTERVENTIONS:
Other: Animal protein based diet
  Arms: Animal protein based diet
Other: Low-nucleotide mycoprotein based diet
  Arms: Low-nucleotide mycoprotein based diet
Other: High-nucleotide mycoprotein based diet
  Arms: High-nucleotide mycoprotein based diet

SUMMARY:
Compare chronic (one week) of a 'normal' meat diet with one week of mycoprotein consumption, with or without a reduced nucleotide content, on markers of metabolic health, such as uric acid concentrations, blood glucose control and blood lipid profiles.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 30

Exclusion Criteria:

* On medication (except contraception)
* Smokers
* Diagnosed with any metabolic or cardiovascular conditions
* BMI < 18 or > 30
* Dietary restrictions (vegetarians/vegans, etc.)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Serum uric acid concentrations | Measured at baseline; days 2, 4 and 6 of the intervention; and after the 1 week intervention (day 8)

SECONDARY OUTCOMES:
Glycaemia and serum insulin - insulin sensitivity (oral glucose tolerance test) | Measured at baseline and after 1 week intervention (day 8)
IL-6 | Measured at baseline and after 1 week intervention (day 8)
24 h blood glucose homeostasis - measured using a Dexcom CGMS | Measured 5 days at baseline (habitual data) and 5 days during the intervention (days 3 - 7)
Metabolomics (using Nuclear Magnetic Resonance - NMR) | Measured at baseline; days 2, 4 and 6 of the intervention; and after the 1 week intervention (day 8)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coelho MOC, Monteyne AJ, Kamalanathan ID, Najdanovic-Visak V, Finnigan TJA, Stephens FB, Wall BT. High dietary nucleotide consumption for one week increases circulating uric acid concentrations but does not compromise metabolic health: A randomised controlled trial. Clin Nutr ESPEN. 2022 Jun;49:40-52. doi: 10.1016/j.clnesp.2022.04.022. Epub 2022 Apr 25. PMID 35623844